CLINICAL TRIAL: NCT01452828
Title: A Phase I Open-Label Study With 200 mg Intravenous TR-701 Free Acid to Assess Safety and Pharmacokinetics in Advanced Renal Impairment Subjects
Brief Title: A Pharmacokinetics and Safety Study in Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Trius Therapeutics LLC, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1986-031; TR701-123 (Other: TriusRX Unique ID)
Record Dates: First submitted 2011-09-21; First posted 2011-10-17 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Renal Impairment
Keywords: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — tedizolid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Renal Impairment Nondialyzed (Experimental)
  Interventions: Drug: TR-701 FA single infusion
- Renal Impairment Dialyzed (Experimental)
  Interventions: Drug: TR-701 FA
- Matched Control (Experimental)
  Interventions: Drug: TR-701 FA

INTERVENTIONS:
Drug: TR-701 FA single infusion — Single IV infusion, 200 mg daily for 7 days
  Other Names: Tedizolid
  Arms: Renal Impairment Nondialyzed
Drug: TR-701 FA — Two separate infusions of 200 mg
  Other Names: Tedizolid
  Arms: Renal Impairment Dialyzed
Drug: TR-701 FA — Single IV infusion, 200 mg daily for 7 days
  Other Names: Tedizolid
  Arms: Matched Control

SUMMARY:
The purpose of this study is to assess the single dose pharmacokinetics (PK) and safety of TR701 FA in subjects with advance renal impairment.

DETAILED DESCRIPTION:
To assess the pharmacokinetics (PK) and evaluate the safety of intravenous (IV) infusion of TR-701 free acid (FA) in subjects with advanced renal impairment compared with matched control subjects with normal renal function

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18.0 and 40.0 kg/m2 inclusive
* Male or female subjects between 18 and 75 years of age
* Stable dosage of medication for 30 days
* for dialysis patients, receiving chronic and stable maintenance hemodialysis for at least 3 months

Exclusion Criteria:

* Functioning transplanted solid organ
* High tyramine diet
* Significant, unstable, or life-threatening condition or organ or system condition or disease, other than kidney disease in renal subjects

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-10; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Composite (or Profile) of Pharmacokinetics | predose, 0.5, 1, 1.5, 2, 2.5, 3, 3.5, 4, 5, 6, 8, 12, 24, 36, 48, 60, 72 hours post-dose
  Cmax, Area Under Curve, Tmax t1/2 will be compared between each renal group and the control group, including calculation of geometric mean ratio and corresponding 90% confidence intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Prokocimer, MD, Study Chair — Trius Therapeutics
Locations (2):
- United States (2):
  - Trius Investigator Site 001, Orlando, Florida
  - Trius Investigator Site 002, Minneapolis, Minnesota

REFERENCES:
- [Derived] Flanagan S, Minassian SL, Morris D, Ponnuraj R, Marbury TC, Alcorn HW, Fang E, Prokocimer P. Pharmacokinetics of tedizolid in subjects with renal or hepatic impairment. Antimicrob Agents Chemother. 2014 Nov;58(11):6471-6. doi: 10.1128/AAC.03431-14. Epub 2014 Aug 18. PMID 25136024